CLINICAL TRIAL: NCT00509509
Title: High Risk Breast Cancer Screening Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Organisation for Oncology and Translational Research (Other)
Other Study IDs: OOTR-SBR001
Record Dates: First submitted 2007-07-29; First posted 2007-07-31 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: Hereditary Breast Cancer (BRCA1, BRCA2)
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer, Familial; Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objectives:

* To screen population with high risk for breast cancer
* To promote the concept and importance of surveillance mammography
* To find out the incidence of breast cancer in population who are in high risk for breast cancer
* To collect blood samples for molecular analysis

ELIGIBILITY:
Inclusion Criteria:

* Female
* > 40 years of age
* Women who have first-degree relative suffered from breast cancer
* Women who have first-degree relative suffered from ovarian cancer
* Family history of male breast cancer
* Family history of breast cancer (not necessarily first degree relatives) diagnosed before age of 40
* Family history of breast cancer (not necessarily first degree relatives) affecting 2 or more family members
* Personal history of ovarian cancer
* Personal history of premalignant conditions of breast and ovary

Exclusion Criteria:

* Women with mammogram within one year

Min Age: 41 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women aged over 40 with high risk of breast cancer
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Louis WC Chow, Principal Investigator — UNIMED Medical Institute
Locations (1):
- UNIMED Medical Institute, Wan Chai, Hong Kong